CLINICAL TRIAL: NCT06057051
Title: A Prospective, Multicenter Study of the Glaukos® iStent Infinite Trabecular Micro-Bypass System Model iS3 in Subjects With Mild to Moderate Primary Open-angle Glaucoma
Brief Title: Glaukos® iStent Infinite Trabecular Micro-Bypass System in Subjects With Mild to Moderate Primary Open-angle Glaucoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLK-401-01
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- iStent Infinite (Experimental): iStent Infinite Trabecular Micro-Bypass System
  Interventions: Device: iStent Infinite

INTERVENTIONS:
Device: iStent Infinite — iStent Infinite Trabecular Micro-Bypass System

SUMMARY:
Prospective, multicenter, single-arm study of the iStent infinite in adult pseudophakic or phakic subjects with mild to moderate primary open angle glaucoma who have not failed conventional medical and surgical treatment

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open-angle glaucoma
* Phakic or pseudophakic
* Age 35 years or older

Exclusion Criteria:

* Traumatic, uveitic, neovascular, angle-closure glaucoma or
* glaucoma associated with vascular disorders
* Active corneal inflammation or edema
* Retinal disorders not associated with glaucoma

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Mean Diurnal Intraocular Pressure (IOP) 12-Month reduction ≥ 20% from Baseline | 12 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Glaukos Investigator Site, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No